CLINICAL TRIAL: NCT07255105
Title: The First Phase of the Closed-loop Improvement Project for Preventing CLABSI
Brief Title: Epidemiological Investigation of Central Venous Catheter-related Bloodstream Infections in Icus in China
Status: Recruiting | Type: Observational
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, Professor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: 2024ZDSYLL338-P01
Record Dates: First submitted 2025-11-16; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: CLABSI - Central Line Associated Bloodstream Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, with the rapid advancement of medical technology and the rapid development of critical care medicine, the use of various central venous catheters in icus has been increasing day by day. Central venous catheter-related bloodstream infection (CLABSI), as a common catheter complication, preventable nosocomial acquired infections have gradually become a focus of attention in the ICU. Once CLABSI occurs, it often leads to a mortality rate as high as 28% to 30% for patients. Data from our country shows that patients with CLASBI will have their hospital stay extended by 8 to 13 days. The additional cost has increased by 3,500 US dollars.

Therefore, over the years, medical systems both at home and abroad have been committed to the prevention and control of CLABSI. The incidence of CLABSI in icus in the United States in 2020 was 0.87 per thousand catheter days. In 2018, the incidence rate of CLABSI in 79 icus in China was 1.5 per thousand catheter days. All the above incidence rates have decreased significantly compared with previous data.

During the COVID-19 pandemic in 2020, the global healthcare system faced severe challenges. Particularly, factors such as the aggravation of patients' conditions in icus, the sharp increase in the use of central venous catheters, the shortage of medical staff, and the ineffective implementation of CLABSI prevention measures jointly led to a significant increase in the incidence of CLABSI. The number of CLABSI cases recorded by the US NHSN in the fourth quarter increased by as much as 47%. In response to this crisis, international and domestic authoritative institutions responded promptly: In 2022, the American Society of Epidemiology (SHEA) updated its prevention strategy for CLABSI. In the same year, the National Health Commission of China emphasized in its medical quality improvement goals the need to reduce intravascular catheter-related infections, especially in the field of critical care medicine, and explicitly indicated the need to lower the incidence of CLABSI in icus.

However, at present, there is still no large-scale investigation on the incidence of CLABSI after COVID-19 in Chinese mainland. This is related to the fact that there is no standard data collection and monitoring platform at present, and the judgment standards and capabilities of various medical institutions are inconsistent.

This study took adult patients with central venous catheters in icus across the country as the research subjects. Through a prospective cohort study, the current incidence and related influencing factors of CLABSI were clarified. To provide a basis and reference for further formulating and implementing CLBASI prevention strategies in the future.

ELIGIBILITY:
Inclusion Criteria:

* 1. Admitted to the ICU with a central venous catheter placed in place and the expected indwelling time exceeds 48 hours (including newly placed central venous catheters or the continued indwelling of existing qualified central venous catheters)

  2. Patients aged 18 or above

  3. Sign the informed consent form

Exclusion Criteria:

1. Patients who have had a central venous catheter indwelled for more than 24 hours before being admitted to the ICU (and are not going to have it replaced immediately)
2. Patients who were re-admitted to the ICU during the study period
3. Lactating and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a central venous catheter in the ICU expected to be retained for more than 48 hours
Sampling Method: Probability Sample
Enrollment: 1846 (Estimated)
Dates: Start 2025-06-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of central venous catheter-related bloodstream infections | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
In the later stage, based on the progress of the research and the actual situation, it will be determined

REFERENCES:
- See also: Online data reporting system — https://cmcr.meddatas.com/